CLINICAL TRIAL: NCT05002946
Title: Phase 1, Open Label, Randomized, Single-dose, 3-Period, 3-Treatment Crossover Study to Evaluate the Pharmacokinetics of SP-104 Under Fasting and Fed Conditions and to Compare to Naltrexone Hydrochloride Tablets USP in Healthy Adult Subjects
Brief Title: Pharmacokinetics of SP-104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SP-104-01
Record Dates: First submitted 2021-08-05; First posted 2021-08-12 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Healthy
MeSH Terms: interventions — Dronabinol; Naltrexone; Tablets

STUDY DESIGN:
Intervention Model Description: Subjects randomized to Treatment A will fast at least 10 hours prior to and for at least 4 hours following dosing and will be treated with a single dose of SP-104. Subjects randomized to Treatment B will be fed a high-fat breakfast 30 minutes prior to dosing, SP-104 will be administered 30 minutes after start of the meal. No food will be allowed for at least 4 hours after the dose. Subjects randomized to Treatment C will fast at least 10 hours prior to and for at least 4 hours following dosing and will be treated with a single dose of Naltrexone Hydrochloride Tablet. Subjects will crossover to each treatment after a wash out period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- A: SP-104 Fasting (Experimental): Oral administration of SP-104 under fasting conditions
  Interventions: Drug: SP-104
- B: SP-104 Under Fed Conditions (Experimental): Oral administration of SP-104 under fed conditions
  Interventions: Drug: SP-104
- Naltrexone Hydrochloride Tablets Fasting (Active Comparator): Oral administration of Naltrexone Hydrochloride Tablets, 50 mg USP under fasting
  Interventions: Drug: Naltrexone Hydrochloride 50Mg Oral Tablet

INTERVENTIONS:
Drug: SP-104 — single oral dose
  Arms: A: SP-104 Fasting; B: SP-104 Under Fed Conditions
Drug: Naltrexone Hydrochloride 50Mg Oral Tablet — single oral dose
  Arms: Naltrexone Hydrochloride Tablets Fasting

SUMMARY:
This open-label, 3-period, 3-treatment, randomized study will characterize the pharmacokinetics and safety and tolerability of SP-104 under fasting and fed conditions as compared to the pharmacokinetics of Naltrexone Hydrochloride Tablets, USP, 50 mg in healthy adult subjects.

DETAILED DESCRIPTION:
The study will characterize the single-dose pharmacokinetics of naltrexone and metabolite (6 Beta-naltrexol) following administration of SP-104 compared to Naltrexone Hydrochloride Tablets, USP, 50 mg in healthy adult subjects under fasting conditions. The study will also characterize the effect of food intake on the pharmacokinetics of SP-104 in healthy adult subjects. Additionally, the safety and tolerability of single doses of SP-104 under fed and fasting conditions will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent , can understand and comply with the requirements of the study, and are able to communicate with the investigator.
* male and female adult subjects between 18 and 65 years.
* Body mass index (BMI) of 18-32 kg/m2.
* Medically healthy
* Agree to total abstinence from heterosexual intercourse, from screening through until at least 30 days after the last study dose, or to the use of an effective method of contraception from screening through until at least 30 days after the last study dose.
* Able to swallow capsules and tablets.

Exclusion Criteria:

* Subject has a history of clinically significant disease, including cardiovascular, GI, renal, hepatic, pulmonary, endocrine, hematologic, vascular, immunologic, metabolic, or collagen disease.
* History of drug or alcohol abuse or dependence based on the DSM-IV criteria as reported by the subject or known to the Investigator.
* Subjects currently dependent on opioids, including those currently maintained on opiate agonists or partial agonists.
* Subjects in acute opioid withdrawal.
* Use of any other investigational drug within 30 days or 6 half-lives, whichever is longer, prior to Day 1 of Period 1.
* Use of prescription medications including opioids, or natural food supplements, alcohol, grapefruit juice, or caffeine within study-specified timeframes.
* Positive urine drug screen for alcohol and drugs of abuse.
* History of allergic or adverse response to naltrexone.
* Serology positive for hepatitis B surface antigen, hepatitis C antibodies, or HIV antibodies.
* Subjects with current or past SARS-CoV-2 infection.
* Are smokers, 'and any use of other types of tobacco or nicotine products within six months prior to Day 1 of Period 1.
* Have donated plasma within 7 days prior Day 1 of Period 1.
* Have donated or lost whole blood prior to administration of the study medication as follows: 50 to 499 mL of whole blood within 30 days, or more than 499 mL of whole within the last 56 days prior to drug administration.
* Have had a serious illness in the 4 weeks preceding the Screening Visit that resulted in missed work or hospitalization (note: subjects missing work due to non-serious illness is not excluded).
* Acute illness, especially any infection, within 4 weeks prior to Day 1 of Period 1.
* Subjects with GFR <90 mL/min at Screening .
* Subjects with any elevation of liver function tests .
* Hemoglobin <12.0 g/dL for males or <10.0 g/dL for females .
* Subjects with a CK value of greater than the upper limit of normal that is not explainable by exercise and that does not come back to reference range upon retest.
* Any history of cancer or any active malignancy except for successfully treated basal cell carcinoma or squamous cell carcinoma.
* Subjects with reported history of, or current treatment for, GI disease such as diverticulitis, diverticulosis, irritable bowel diseases, ulcer, inflammatory bowel disease or history of conditions, such as abdominal gunshot wounds.
* Are an employee, family member, Sponsor, or student of the Investigator or of the clinical site.
* Clinical judgment by the investigator that the subject should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-04-24 (Actual)

PRIMARY OUTCOMES:
Concentration of SP-104 | 72 hours
  Observed plasma concentrations of naltrexone and metabolite 6β-naltrexol ng/mL
Time to maximum concentration of naltrexone and metabolite 6β-naltrexol | 72 hours
  Time to maximum plasma concentration of naltrexone and metabolite 6β-naltrexol in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, MD, Study Director — Scilex Pharmaceuticals, Inc.
Locations (1):
- Christchurch Clinical Studies Trust (NZCR), Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No